CLINICAL TRIAL: NCT00721747
Title: Phase II, Open, Not Randomized Clinical Trial, to Evaluate the Sequential Taxotere®, Followed by Myocet® and Cyclophosphamide First Line Treatment in her2 Negative Breast Cancer Patients
Brief Title: Taxotere®, Followed by Myocet® and Cyclophosphamide First Line Treatment in HER2 Neg Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Oncológico Gallego (Other)
Collaborators: Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG/2007-01; 2007-005173-56
Record Dates: First submitted 2008-07-23; First posted 2008-07-24 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: breast cancer patients her2 negative pathological responses
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Unique arm (Experimental): 4 cycles of Docetaxel 100mg/m2 iv followed by 4 cycles of Liposomal doxorubicine 60mg/m2/iv and Cyclophosphamide 600mg/m2/iv
  Interventions: Drug: Docetaxel, Liposomal doxorubicine and Cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel, Liposomal doxorubicine and Cyclophosphamide — 4 cycles of Docetaxel 100mg/m2 iv followed by 4 cycles of Liposomal doxorubicine 60mg/m2/iv and Cyclophosphamide 600mg/m2/iv

SUMMARY:
The purpose of this study is to determine how many pathological complete responses are achieved in patients treated with taxotere® (T) followed by Myocet® (M)and Cyclophosphamide (MC) first line treatment in HER2 negative brest cancer patients.

DETAILED DESCRIPTION:
Phase II, open, not randomized clinical trial, to evaluate the sequential Taxotere®, followed by Myocet® and Cyclophosphamide first line treatment in her2 negative breast cancer patients.

The purpose of this study is to determine how many pathological complete responses are achieved in patients treated with taxotere® (T) followed by Myocet® (M)and Cyclophosphamide (MC) first line treatment in HER2 negative brest cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Brest adenocarcinoma stages II/III
* Female
* Informed consent signed
* HER2 negative
* Age>18 years old
* ECOG < 1
* Proper organic function regarding the following criteria:

  1. ANC > 2,0 x 109L, platelets > 100 x 109L and hemoglobin > 10g/dL (transfusion is allowed)
  2. Hepatic Function:

  i.Bilirubin < 1,5 x UNL ii.AST ,ALT < 2,5 x UNL iii.Alkaline phosphatase < 5 UNL iv.Patients with AST and /or ALT > 1.5 x UNL and alkaline phosphatase > 2.5 x UNL will not be selected for the study c.Renal function: creatinine < 1,25 x UNL, or creatinine clearance > 60 mL/min d.Normal Cardiac function, confirmed with FEVI >50% and electrocardiogram.
* Patients should be available for treatment and follow up and must be treated in investigator or co-investigator site
* Negative pregnancy test(performed 7 days before treatment)

Exclusion Criteria:

* Previous treatment for breast cancer (CT, RT, IT, HT)
* Stages IIIb, IIIc or IV or invasive bilateral breast cancer
* Previous neoplasias treated with Anthracyclines or Taxanes (Paclitaxel or Docetaxel)
* Pregnant or breastfeeding females
* Neurotoxicity Grade 2
* FEV≤50% or any cardiac disease in which anthracyclines are contraindicated
* Other severe diseases regarding investigator criteria
* Any neurological or psychiatric pathology
* Previous neoplasia different from breast cancer except:

  1. skin cancer(no melanoma)
  2. In situ cervix Carcinoma
  3. Ipsilateral in situ ductal carcinoma
  4. In situ lobular in situ carcinoma
  5. Any other carcinoma without evidence disease in last 10 years
* Treatment chronic with corticoids (except patients starting 6 months before inclusion with low dosages (* 20 mg methylprednisolone or equivalent)
* Concomitant treatment with Hormone ovarian replacement therapy
* Contraindication for corticoids
* Concomitant treatment with another investigational drugs
* Included in another clinical trial with any drug in 30 days before inclusion study
* Concomitant treatment with another anticancer therapy
* Male patients
* Hypersensibility to any study drug or components

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Determine proportion of Pathological complete responses | At the end of the treatment, after Surgery.

SECONDARY OUTCOMES:
Determine proportion of clinical responses | At the end of the treatment
Describe treatment safety | At the end of the treatment
Determine proportion of conservative breast surgery | At the end of the study
Evaluate disease free survival | At the end of the treatment
Evaluate Overall survival | At the end of the treatment
Evaluate gene patterns regarding prediction of treatment response | At the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jesús García Mata, MD, Principal Investigator — Grupo Oncológico Gallego
Locations (6):
- Spain (6):
  - Hospital de Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Juan Canalejo, A Coruña, Galicia
  - Centro Oncológico de Galicia, A Coruña, Galicia
  - Complejo Hospitalario de Ourense, Ourense, Galicia
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Xeral Cies, Vigo, Galicia